CLINICAL TRIAL: NCT03130218
Title: Aromatherapy in Management of Postoperative Nausea in Post-Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-74-LGH
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Bariatric Surgery Candidate; Nausea, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Randomized by day of week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control group will not receive peppermint oil aromatherapy as a primary intervention for postoperative nausea and vomiting. Primary therapy for postoperative nausea and vomiting would entail standard antiemetic drug therapies. Patient monitoring and documentation would include the following: Patients in the control group will be assessed every 4 hours and as needed for nausea. All aspects of care from physician, nursing and all disciplines will be consistent with current practices in care of postoperative bariatric surgical patients.
- Intervention (Experimental): Patients in the intervention group will receive peppermint oil aromatherapy as primary treatment for postoperative nausea. Pharmacological therapy with anti-nausea drug therapies will be available as needed. All other aspects of medical, surgical and nursing care will be standard practice for pre and post-operative care related to the bariatric surgical patient. Patients in the intervention group will be assessed every 4 hours and as needed for nausea. Post-intervention, the patient will be re-assessed for level of nausea after one hour. In the event the patient refuses peppermint oil aromatherapy and requests anti-emetic drug therapies, they are able to do so.
  Interventions: Other: Peppermint oil aromatherapy

INTERVENTIONS:
Other: Peppermint oil aromatherapy — Aroma therapy with peppermint oil administered with presoaked diffuser and bag.
  Arms: Intervention

SUMMARY:
Determine the effectiveness of peppermint oil aromatherapy in relieving post-operative nausea in the bariatric surgery patient population.

DETAILED DESCRIPTION:
Healthy weight management and use of essential oils and aromatherapy as natural interventions to manage health-related issues are significantly growing interests. One frequent intervention for healthy weight management is bariatric surgery. In the post-operative period following bariatric surgery, nausea is a common consequence. Peppermint oil aromatherapy is an effective intervention for relieving nausea and other gastrointestinal symptoms in the bariatric and surgical population. This study has multiple aims. One is to determine effectiveness of peppermint oil aromatherapy in relieving post-operative nausea in the bariatric surgery patient population. A second aim is to establish relative cost-effectiveness of peppermint oil aromatherapy versus traditional anti-emetic drug therapies. A third is to determine whether peppermint oil aromatherapy increases patient satisfaction versus anti-emetic drug therapies. This is a randomized study with control and experimental groups. The control group will receive no peppermint oil aromatherapy and only traditional anti-emetics as needed. The experimental group will receive peppermint oil aromatherapy and traditional anti-emetics as needed.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery candidate on 7-Lime at Lancaster General Hospital
* Scheduled for laparoscopic sleeve gastrectomy and laparoscopic Roux-En-Y (RNY) procedures
* Between ages of 18 and 70
* Surgical patient of either Dr. James Ku and Dr. Joseph McPhee

Exclusion Criteria:

* History of excessive sensitivity to peppermint oil, allergic response to peppermint oil and who state preference against aromatherapy
* Not alert and oriented or unable to follow directions will be excluded
* Severe reactive airway disease such as asthma or chronic obstructive pulmonary disease (COPD)
* Possible exclusion for severe hypertension or atrial fibrillation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Nausea Assessment and Treatment Scale | 4 Hours
  Severity of post-operative nausea on a scale of 0-10
Count of Antiemetic Drug Therapies | 4 Hours
  Number of antiemetic drug therapies used in the post-operative period
Perception of Postoperative Nausea Management Survey | 24 Hours
  Patient satisfaction with effectiveness of postoperative nausea management

CONTACTS AND LOCATIONS:
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson LA, Gross JB. Aromatherapy with peppermint, isopropyl alcohol, or placebo is equally effective in relieving postoperative nausea. J Perianesth Nurs. 2004 Feb;19(1):29-35. doi: 10.1016/j.jopan.2003.11.001. PMID 14770380
- [Background] Tate S. Peppermint oil: a treatment for postoperative nausea. J Adv Nurs. 1997 Sep;26(3):543-9. doi: 10.1046/j.1365-2648.1997.t01-15-00999.x. PMID 9378876
- [Background] Lane B, Cannella K, Bowen C, Copelan D, Nteff G, Barnes K, Poudevigne M, Lawson J. Examination of the effectiveness of peppermint aromatherapy on nausea in women post C-section. J Holist Nurs. 2012 Jun;30(2):90-104; quiz 105-6. doi: 10.1177/0898010111423419. Epub 2011 Oct 27. PMID 22034523